CLINICAL TRIAL: NCT01394302
Title: Functional Profile of People Suffering From Trigger Finger
Brief Title: The Functional Profile of People Suffering From Trigger Finger
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Dr Michaeil Michaeilovich - Sheruty Briut Clalit, Dr Michaeil Michaeilovich - Sheruty Briut Clalit
Other Study IDs: 054/2011ק
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-06

CONDITIONS: Trigger Finger
Keywords: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to Characterize the population of people who suffer from trigger finger (TF) in terms of demographic (Gender, age, occupation, etc.); motor skills (hand function); the Consequences of the disease on a person's daily functioning and impact on quality of life.

The study will also attempt to examine the suitability of several common assessment tool for evaluation of hand rehabilitation Patients who suffer from TF.

Information obtained from the study will enable a deeper comprehension of the consequences of TF on the patient and will be the first step in developing a protocol assessment and evidence-based treatment in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 and above.
* Men and Women.
* diagnosed with Trigger Finger.

Exclusion Criteria:

* Trauma in upper Extremity.
* Cognitive difficulties that are blocking the ability to answer the questionnaires (dementia, head injury).
* Pregnant women.
* participants who didnt completed all Assessments.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who come to visit The hand Specialist doctor and receive a diagnosis of TF.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michaeil Michaeilovich, M.D., Principal Investigator — Sherutey Briut Clalit
Locations (1):
- Sherutey Briut Clalit, Jerusalem, Israel